CLINICAL TRIAL: NCT05059834
Title: Feasibility and Acceptability of an Evidence-based Mindfulness Online Resources for Patients With Generalized Anxiety Disorder
Brief Title: Feasibility Study for Online Mindfulness for GAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.385
Record Dates: First submitted 2021-09-13; First posted 2021-09-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Anxiety Generalized
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- online mindfulness resources + usual care (Experimental): The mindfulness online resources consisted of 4 weekly modules. Mindfulness exercises, including body scan, mindful breathing, mindful eating, mindful walking, 3-min breathing space, and thought distancing exercise, are audio-recorded to facilitate participants to practice mindfulness. Readings and graphics are included to explain the concept of mindfulness and to share with participants the common difficulties that participants may come across during mindfulness practices.
  Interventions: Behavioral: online mindfulness resources
- usual care (Other): patients will receive usual care from doctors
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: online mindfulness resources — a free mindfulness resource online for patients with general anxiety disorder
  Arms: online mindfulness resources + usual care
Behavioral: usual care — patient will continue to receive drug and advice from doctors and nurses for their anxiety disorder
  Arms: usual care

SUMMARY:
Method: . Forty patients with general anxiety disorder will be randomized in 1:1 ratio to the online resource plus usual care, and to usual care control group by stratified block randomization. Measurements including 7-item Generalized Anxiety Disorder questionnaire, 9-item Patient Health Questionnaire, Penn State Worry questionnaire, and Five Facet Mindfulness Questionnaire will be made at baseline and at 2-month. Rate of recruitment, drop out and website usage will be collected. All patients in the intervention arm will be interviewed to assess the clarity of the app and user experience. The scores between the two arms will be compared by t-test and the transcripts of the patient interviews will be analysed using thematic analysis

ELIGIBILITY:
Inclusion Criteria:

* received a diagnosis of GAD in the computerized record system (CMS) in Hong Kong hospital authority
* score ≥10 on the 7-item Generalized Anxiety Disorder scale (GAD-7), signifying active moderate anxiety symptoms
* used any website in prior 12 months
* received stable dose of psychoactive medications in last 2 months

Exclusion Criteria:

* any diagnosed psychotic disorder
* diagnosis of dementia
* any diagnosed substance abuse disorder (except smoking)
* active suicidal ideation (score ≥1 on 9-item Patient Health Questionnaire
* had regular mindfulness meditation practice in last 6 months or had participated in MBSR/MBCT course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
recruitment rate | through study completion, an average of 1 year
  rate of recruitment during the trial period
dropout rate | through study completion, an average of 1 year
  rate of dropout during the trial period

SECONDARY OUTCOMES:
7-item Generalized Anxiety Disorder questionnaire | baseline and 2-month
  a validated questionnaire to measure anxiety symptoms. Possible score ranged from 0-21. the higher the score, the more severe the anxiety symptoms
9-item Patient Health Questionnaire | baseline and 2-month
  a validated questionnaire to measure anxiety symptoms. Possible score ranged from 0-27. the higher the score, the more severe the depressive symptoms
Penn State Worry Questionnaire | baseline and 2-month
  a validated questionnaire to measure worry. The possible score ranged from 16-80. the higher the score, the more severe the worries
Five Facet Mindfulness Questionnaire | baseline and 2-month
  a validated questionnaire to measure mindfulness. The possible score ranged from 1-5. the higher the score, the more mindful the participants are

CONTACTS AND LOCATIONS:
Locations (1):
- School of public health and primary care, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
will share on a reasonable request from other researchers